CLINICAL TRIAL: NCT00387582
Title: Lucentis in the Treatment of Macular Edema - A Phase II, Single Center, Randomized Study to Evaluate the Efficacy of Ranibizumab Versus Focal Laser Treatment in Subjects With Diabetic Macular Edema
Brief Title: Efficacy Study of Lucentis in the Treatment of Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rocky Mountain Retina Consultants (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Roy A. Goodart, M.D., Principal Investigator, Rocky Mountain Retina Consultants
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF3799S
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
Keywords: Diabetes; Macular Edema; Diabetic Retinopathy; Lucentis; Ranibizumab
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Macular Edema | interventions — Ranibizumab; Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Lucentis injections for the first three months of the study and then per the protocol for the duration of the trial.
  Interventions: Drug: Ranibizumab (Lucentis)
- II (Active Comparator): Argon Laser treatment at enrollment and then per the protocol for the duration of the study.
  Interventions: Procedure: Argon Laser

INTERVENTIONS:
Drug: Ranibizumab (Lucentis) — Lucentis 0.5 mg monthly for the first three months and then per protocol for the duration of the trial.
  Other Names: NDC # 50242-0080-01, Brand Name is Lucentis
  Arms: I
Procedure: Argon Laser — Argon laser at entry to trial and then per protocol for the duration of the study.
  Arms: II

SUMMARY:
This study will evaluate the clinical efficacy of intra-vitreal injections of Ranibizumab (Lucentis) in the treatment of Diabetic Macular Edema as compared to grid/focal laser.

DETAILED DESCRIPTION:
Diabetic macular edema (DME) results from abnormal leakage of macromolecules into the extracellular space from microaneurysms and incompetent blood vessel walls due to small vessel damage from high blood glucose levels. Oncotic forces then allow water into the extracellular space. Abnormalities in the retinal pigment epithelium (RPE) may reduce normal outflow of fluid from the retina to the underlying choriocapillaris via the pump mechanism (Ferris et al. 1984). This leads to retinal edema in the macula with accompanying loss of vision. There is evidence suggesting that vascular endothelial growth factor (VEGF) plays a part in vessel wall permeability with subsequent retinal edema (Aiello et al. 1997).

Studies demonstrate that tight junctions in the vessel walls were shown to be regulated by VEGF and VEGF increases vascular permeability (Anticliff et al. 1999). The healthy human retina contains little or no VEGF. Hypoxia, a component of diabetic retinopathy, causes upregulation of VEGF in the retina (Vinores et al. 1997). Binding VEGF with an antibody specific for VEGF may inhibit resultant edema thus preventing and possibly reversing loss of vision.

Diabetic retinopathy is the leading cause of blindness in people aged 20-74 years, accounting for 8% of all cases of legal blindness and 12% of the newly blind (Klein 1995). A common complication of all forms of diabetes mellitus, diabetic retinopathy is present in over 2.5% of the U.S. population, or more than 5.3 million people aged 18 or older (Prevent Blindness American 2002).

Three forms of retinopathy are commonly recognized in association with all forms of diabetes mellitus: 1) non-proliferative diabetic retinopathy (NPDR), 2) proliferative diabetic retinopathy (PDR), and 3) diabetic macular edema (DME).

NPDR is characterized by ophthalmoscopically visable abnormalities that include microaneurysms, intraretinal hemorrhages, exudates, retina nerve fiber layer infarcts (cotton-wool spots), and, in more severe cases, venous beading and intraretinal microvascular abnormalities (IRMA).

Over time, NPDR may progress to more severe PDR, the hallmark of which is neovascularization on the surface of the retina, optic disc, or iris, and angle structures in the front of the eye. PDR is associated with a high risk of visual morbidity arising from vitreous hemorrhage, traction retinal detachment, and neovascular glaucoma (Diabetic Retinopathy Research Group 1979).

DME, the third form of diabetic retinopathy, is characterized by swelling of the central part of the retina that mediates high-resolution vision. DME frequently coexists with and is superimposed upon NPDR or PDR. When the area of swelling is located more than 1 disc diameter (approximately 1500 mm) away from the center of the fovea, the swelling constitutes a low threat to visual acuity and is regarded as non-clinically significant macular edema (Early Treatment Diabetic Retinopathy Study [ETDRS] Research Group 1985). Vision deteriorates when DME involves the foveal center. DME that either directly involves the fovea or is at high risk of doing so is referred to as Clinically Significant Macular Edema (CSME) (ETDRS Research Group 1985).

When the center of the fovea is involved by CSME, the DME is referred to as CSME with center involvement (CSME-CI), as opposed to CSME without center involvement (ETDRS Research Group 1987).

The natural history of untreated CSME-CI is particularly poor. The ETDRS demonstrated that over a 3-year period, 33% of subjects with CSME-CI lose >15 letters of visual acuity on the standardized ETDRS Visual Acuity Chart (Ferris et al. 1982) compared with 23% of CSME subjects without center involvement (ETDRS Research Group 1987). Such a degree of visual acuity change is equivalent to doubling of the visual angle or greater. The ETDRS did not discriminate between subtypes of diabetes mellitus.

Although laser photocoagulation in CSME-CI was shown to reduce the proportion of subjects losing > 15 letters from 33% to 13% over 3 years, 13% of subjects nevertheless continued to double their visual angle or do worse. Moreover, in subjects with CSME initially without center involvement, over 3 years, 12% lose > 15 letters despite laser treatment, presumably because edema eventually involves the center of the fovea (i.e., the subjects convert to CSME-CI). Thus, while laser is an effective tool in the treatment of CSME, there is a considerable unmet clinical need for CSME-CI.

This study is designed to compare the effectiveness of intra-vitreal Ranibizumab to current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:

  * Clinically significant diabetic macular edema (CSME) or clinically significant diabetic macular edema with center involvement (CSME-CI) as defined by the ETDRS Trial (ETDRS Research Group 1987 and 1991)
  * Retinal thickening within 500 mm of the center of the fovea
  * Hard exudates within 500 mm of the center of the fovea (if associated with adjacent retinal thickening, which may be outside of 500um limit)
  * An area of macular edema greater than 1 disc area but within 1 disc diameter of the center of the macula
  * Ability to provide written informed consent and comply with study assessments for the full duration of the study
  * Age > 21 years
  * Visual acuity < 20/320 with definite retinal thickening due to diabetic macular edema based on clinical exam
  * Retinal thickness on OCT measuring 250 microns or more in the central subfield or 350 microns of more in any non-central subfield
  * Media clarity and pupillary dilatation, patient cooperation, and adequate fundus photographs and OCT will be obtainable
  * No other ocular conditions that could cause macular edema will be present

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:

  * Other causes of macular edema will be present
  * Intraocular pressures exceed 25 mm Hg
  * Prior enrollment in the study
  * Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
  * Participation in another simultaneous medical investigation or trial or previous trial of Lucentis or Avastin
  * Premenopausal women not using adequate contraception The following are considered effective means of contraception: surgical sterilization, use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch
  * Pregnancy or lactation (evidenced by Early Pregnancy Test (EPT) over the counter test)
  * Current treatment of a systemic infection
  * Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders
  * History of recurrent significant infections or bacterial infections
  * Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either

    * Require medical or surgical intervention during the 12-month study period to prevent or treat visual loss that might result from that condition, or
    * If allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA over the 12-month study period
  * Active intraocular inflammation (grade trace or above) in the study eye
  * Current vitreous hemorrhage in the study eye
  * History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
  * History of idiopathic or autoimmune-associated uveitis in either eye
  * Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
  * Concurrent ocular disease associated with choroidal neovascularization to include but not limited to presumed ocular Histoplasmosis, high myopia, or macular degeneration
  * Prior/Concomitant Treatment
  * Patient will not have had panretinal photocoagulation treatment within 4 months
  * Grid/focal laser within 2 months of randomization
  * Subtenon steroid in study eye within 6 months
  * Treatment with systemic steroid currently or within the last 4 weeks
  * IVTA within 3 months
  * Previous participation in any studies of investigational drugs within 30 days preceding Day 0 (excluding vitamins and minerals)
  * Prior participation in a Genentech ranibizumab clinical trial
  * Previous treatment with intravitreally (in either eye) or intravenously administered Avastin (bevacizumab)
  * Concurrent use of systemic anti-VEGF agents
  * Previous use of Macugen in study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Prevention of vision loss at one year as evidenced by ETDRS visual acuity. | 6 and 12 months

SECONDARY OUTCOMES:
Reduction in retinal thickening based on Optical Coherence Tomography. | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roy A. Goodart, MD, Principal Investigator — Rocky Mountain Retina Consultants
Locations (1):
- Rocky Mountain Retina Consultants, Salt Lake City, Utah, United States